CLINICAL TRIAL: NCT03761290
Title: Glucose Homeostasis and Beta Cell Function in Pseudohypoparathyroidism
Brief Title: Glucose Homeostasis in Pseudohypoparathyroidism
Status: Terminated | Type: Observational
Why Stopped: COVID precautions prevented enrollment of healthy controls, funding ended.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ashley Shoemaker, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: Shoemaker R03
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Pseudohypoparathyroidism and Pseudopseudohypoparathyroidism; Pseudohypoparathyroidism Type Ia; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism; Pseudopseudohypoparathyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pseudphypoparathyroidism type 1A (PHP1A): Case
- Pseudopseudohypoparathyroidism (PPHP): Case
- Controls: Matched control group

SUMMARY:
It is increasingly recognized that Pseudohypoparathyroidism type 1A (PHP1A) is associated with an increased risk of type 2 diabetes but the mechanism is unknown. In this pilot study we will assess β-cell function in patients with PHP1A and pseudopseudohypoparathyroidism PPHP.

DETAILED DESCRIPTION:
Pseudohypoparathyroidism type 1A (PHP1A) is a rare, genetic disorder caused by impaired stimulatory G-protein signaling due to heterozygous mutations in the gene, GNAS. The most severe form of the disease, PHP1A occurs when a GNAS mutation is inherited on the preferentially expressed maternal allele. A less severe form of the disease, pseudopseudohypoparathyroidism (PPHP), occurs when a GNAS mutation is inherited on the paternal allele. Clinically, PHP1A is characterized by multi-hormone resistance, cognitive impairment and early-onset obesity while PPHP has a mild phenotype without multi-hormone resistance. It is increasingly recognized that PHP1A is associated with an increased risk of type 2 diabetes but the mechanism is unknown. Glucose homeostasis and diabetes risk has not been studied in PPHP. As part of the parent K23 award, we investigated glucose tolerance in children with PHP1A. In contrast to the adult literature, we found that children with PHP1A had greater insulin sensitivity than matched controls. When challenged with an oral glucose load, however, children with PHP1A had persistent hyperglycemia and 25% met criteria for impaired glucose tolerance. The goal of this proposal is to quantify β-cell function in PHP1A. It is plausible that these individuals have a) impaired β-cell function, b) differences in insulin sensitivity, and c) impaired incretin function. Thus, in this pilot study we will definitively assess one of these, β-cell function, using the frequently sampled intravenous glucose tolerance test in patients with PHP1A and PPHP (aim 1). We will also assess oral glucose tolerance over time by bringing back children and young adults with PHP1A from our original cohort for repeat glucose tolerance testing (aim 2). The ultimate goal is to rigorously define glucose homeostasis defects in PHP1A in order to design and conduct an intervention study for glucose intolerance and type 2 diabetes in PHP1A.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PHP1A/PPHP
2. Age between 6 and 50 years old

Controls will be matched based on:

1. Gender
2. Race
3. Age (±2 years if <25 years old or ±5 years if ≥25 years old)
4. BMI (±2 kg/m2)
5. Diabetes status

Exclusion Criteria:

1. Treatment with appetite-altering drug or initiation of a new weight loss program in the past 3 months
2. Type 1 diabetes
3. Type 2 diabetes treated with insulin or GLP-1 receptor agonists or A1c >9%at their most recent clinic visit
4. Pregnant or lactating women

Ages: 6 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with PHP1A/PPHP and matched controls
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (Si) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ashley H Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez KM, Curley KL, Slaughter JC, Shoemaker AH. Glucose Homeostasis and Energy Balance in Children With Pseudohypoparathyroidism. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4265-4274. doi: 10.1210/jc.2018-01067. PMID 30085125
- See also: Vanderbilt PHP Research Page — http://www.facebook.com/pseudohypoparathyroidism